CLINICAL TRIAL: NCT06434922
Title: A Randomized Clinical Trial Study on the Prevention Strategy and Early Detection of Ulcer Recurrence in Patients With Type II Diabetes Mellitus Using the Risk of Recurrence Ulcer Tool
Brief Title: Prevention and Early Detection of Ulcer Recurrence in Patients With Type II Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute Technology and Health Muhammadiyah West Kalimantan (Other)
Responsible Party: Principal Investigator, Haryanto Haryanto, Principal Investigator, Institute Technology and Health Muhammadiyah West Kalimantan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ID01
Record Dates: First submitted 2024-05-18; First posted 2024-05-30 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Recurrence; Diabetic Foot; Thermography; Quality of Life
MeSH Terms: conditions — Recurrence; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Intervention group: patient education covered various aspects, including regular monitoring of blood glucose levels, effective dietary management, consistent physical activity, routine foot inspections, adherence to prescribed medications, and appropriate footwear selection based on plantar foot pressure measurements.
  During the intervention procedure, data collection sessions lasted approximately 1 to 1.50 hours, with education and foot care provided once a month. Subsequently, patients underwent monthly follow-ups for three months, during which they received guidance on foot examination, foot care, dietary habits, physical exercise, and stress management.
  Control group: Patients were educated about DM management, medication adherence, dietary practices, physical exercise routines, and foot care through pamphlets.
Masking Description: The investigators known the groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Strategies (Experimental): Groups received the prevention strategies to prevent the recurrence of DFU's
  Interventions: Device: Prevention Strategies
- Standard Strategies (Other): Groups received the standard strategies to prevent the recurrence of DFU's
  Interventions: Device: Standard Strategiies

INTERVENTIONS:
Device: Prevention Strategies — Data collection sessions lasted approximately 1 to 1.50 hours, with education and foot care provided once a month. Subsequently, patients underwent monthly follow-ups for three months, during which they received guidance on foot examination, foot care, dietary habits, physical exercise, and stress management.
  Arms: Prevention Strategies
Device: Standard Strategiies — Group were educated about DM management, medication adherence, dietary practices, physical exercise routines, and foot care through pamphlets
  Arms: Standard Strategies

SUMMARY:
The goal of this clinical trial is to to evaluate the effectiveness of prevention strategies of recurrence in DFU's. It will also to detect the risk level of recurrence. The main question it aims to answer are:

* Does intervention of prevention strategies effective to prevent the recurrence of DFU's?
* How the risk level of the recurrence on DFU's patients?
* How the impact of quality of life on DFU's patients?

Researchers will compare intervention groups (receiving education covered various aspects, including they received guidance on foot examination, foot care, dietary habits, physical exercise, and stress management), and control groups (received standards follow-up care provided by healthcare providers, including pamphlets outlining care for DM patients based on the five pillars, including DM management, medication adherence, dietary practices, physical exercise routines, and foot care).

Participants will:

* For intervention group will be educated every month
* Data for both intervention and control groups were collected monthly until three months.

DETAILED DESCRIPTION:
1. Introduction

   A recurrence of a diabetic foot ulcer refers to the emergence of a new foot ulcer in individuals with a prior history of foot ulceration, irrespective of the specific location or duration since the occurrence of the previous ulcer. Even after the resolution of a foot ulcer, recurrence remains a common problem. In Indonesia, studies have indicated a recurrence rate of diabetic foot ulcers ranging from 13.30% to 35%, while global recurrence rates vary significantly among different countries. Thus, implementing prevention strategies is crucial in averting recurrence. These strategies, such as proper foot care, glycemic control, and early detection and management of risk factors, can significantly reduce the occurrence and recurrence of diabetic foot ulcers.

   Several studies have highlighted various preventive treatments aimed at decreasing the likelihood of diabetic foot ulcer recurrence. These treatments include integrated foot care, self-management techniques, patient education, therapeutic footwear utilization, and surgical intervention. Recent research has also explored the potential of thermography in detecting foot ulcer risk among patients with diabetes mellitus. While numerous original studies and systematic reviews have reported prevention strategies for preventing diabetic foot recurrence, there is limited research on the combined approach of early detection and prevention of foot ulcer recurrence.

   In Indonesia, preventive strategies for diabetes mellitus patients have been implemented through the PROLANIS program, a chronic disease management initiative launched in 2010 in community health centers. PROLANIS focuses on diabetes self-management and follows the five-pillar method established by the Indonesian Society of Endocrinology (PERKENI), encompassing dietary practices, physical activity, pharmaceutical interventions, glucose monitoring, and educational initiatives. Despite the nationwide adoption of these pillars since 2011, the prevalence of recurrence remains significant in Indonesia. Prevention strategies, carried out by healthcare provider teams, including nursing staff, are vital in addressing this challenge. Nurses are involved in physical assessment, early detection, foot care, and education, making their role crucial in implementing prevention strategies.

   Early detection is integral to preventing ulcer recurrence. A systematic review identified three main types of interventions used in early ulcer recurrence detection: conventional physical assessment, 3D thermal camera assessment systems, and diabetic foot screening instruments. Hence, further development of early detection methods for recurrence risk is necessary.

   The study utilized a multifaceted approach incorporating four techniques to reduce the risk of ulcer recurrence in patients with DM. These strategies included:1) conducting a thorough physical examination and assessing the foot, which involved utilizing a thermograph to identify variations in skin temperature; 2) implementing appropriate foot care practices; 3) providing patients with educational resources and guidance; and 4) promptly identifying and addressing factors that may increase the likelihood of ulcer recurrence.

   1.1. Objective The primary objective of this study is to assess the efficacy of preventive measures while ascertaining the degree of risk associated with potential recurrences using the risk of recurrence ulcer tool. Additionally, an assessment was conducted to evaluate the impact on the quality of life.
2. Methods and Materials 2.1. Study Design and Participants This study is prospective clinical trial design to evaluate the effectiveness of prevention strategies utilizing an early detection tool for ulcer recurrence. The study had approved by the ethics committee of the Institute of Technology and Health Muhamamdiyah West Kalimantan. Conducted between January and July 2023 at two community health centers in Pontianak and Kubu Raya, West Kalimantan, Indonesia, the study followed the Consolidated Standards of Reporting Trials (CONSORT); randomized controlled trial (RCT) guidelines principles. Sixty participants were recruited using simple random allocation sampling, with 30 individuals assigned to each group based on calculated sample size requirements. G Power software was utilized to determine sample size, considering a significance level (α) of 0.05, power (β) of 0.95, proportion (p1) of 0.12 in group 1, and proportion (p2) of 0.54 in group 2. Inclusion criteria included the ability to perform everyday tasks, cooperation, and ulcer recovery for at least two weeks, while exclusion criteria comprised serious illnesses or sequelae, active foot ulcers, Charcot neuro-osteoarthropathy, persistent limb-threatening ischemia, and foot infections.

Participants who had received care at the community health centers and had recovered from their wounds constituted the intervention and control groups. Recruitment involved searching medical records and contacting eligible individuals. Written informed consent was obtained before enrollment. The 60 participants were divided into intervention and control groups. Both groups were encouraged to visit the community health centers, with researchers conducting home visits if necessary. The intervention group received the study's treatment, while the control group received standard follow-up care provided by healthcare providers, including pamphlets outlining care for DM patients based on the five pillars, including ulcer prevention.

2.2. Data Collection In this investigation, four research assistants underwent training following the study protocol to conduct examinations on diabetic feet, which included utilizing tools such as the thermograph, monofilament test, vascular Doppler ultrasound, conventional foot plantar scan, and diabetic foot and nail care. Additionally, they were trained in collecting demographic data, assessing diabetic wounds, and educating patients. Patient education covered various aspects, including regular monitoring of blood glucose levels, effective dietary management, consistent physical activity, routine foot inspections, adherence to prescribed medications, and appropriate footwear selection based on plantar foot pressure measurements. Following plantar foot pressure measurement, patients were educated on maintaining regular blood sugar control, dietary management, exercise routines, foot inspection practices, medication adherence, and proper footwear selection.

During the intervention procedure, data collection sessions lasted approximately 1 to 1.50 hours, with education and foot care provided once a month. Subsequently, patients underwent monthly follow-ups for three months, during which they received guidance on foot examination, foot care, dietary habits, physical exercise, and stress management.

For the control group, a comprehensive foot examination was conducted at the initial assessment to evaluate the overall foot health of participants. Patients in the control group were educated about DM management, medication adherence, dietary practices, physical exercise routines, and foot care through pamphlets. Data for both intervention and control groups were collected monthly through examinations and inspections, each conducted by two nurses who had completed preventive foot care training.

Throughout the study, data collection included vascular Doppler ultrasonography (BT-200 V, 8 MHz; Bistos Co., Ltd., Seongna, Korea) for assessing the ankle-brachial index (ABI) and the monofilament test using a 10-g (5.7) Semmes-Weinstein monofilament to evaluate neuropathic status. Additionally, plantar pressure distribution data were collected using a foot printer (Bauerfeind AG, Thuringia, Germany) and a callus removal device. Clinical examinations were conducted to assess structural and functional foot deformities, including claw/hammer toe, hallux rigidus, hallux valgus, bony prominences, pes cavus, pes planus, and metatarsal head abnormalities.

The risk level recurrence ulcer tool, INDIFURUTO (Indonesian Diabetic Foot Ulcer Recurrence Assessment Tool), was utilized to assess the risk level. INDIFURUTO considers factors such as history of amputation, smoking, serum glucose levels, ankle-brachial index, monofilament test results, and differences in foot skin temperature. Skin temperature measurements were obtained using smartphone-based thermography (FLIR ONE Gen 3, Teledyne FLIR LLC, Wilsonville, OR, USA). Subjects were categorized as high risk if they scored less than or equal to 22 points, medium risk if they scored between 23 and 45, and low risk if they scored more than or equal to 46. Previous studies have demonstrated high sensitivity (100%) and specificity (90%) of this tool. INDIFURUTO assessments were conducted at baseline, and at the second and third follow-up assessments for both groups.

The European Quality of Life 5 Dimensions 3 Level (EQ-5D-3L) version was utilized to evaluate participants' quality of life, a measure that has demonstrated reliability with a Cronbach's alpha coefficient of 0.79. Quality of life assessments were conducted at baseline, as well as at the second and third follow-up assessments for both intervention and control groups. Participants self-assessed their level of mobility, self-care, usual activities, pain or discomfort, and anxiety or depression, with responses ranging from level 1 (indicating the best state) to level 3 (indicating the worst state). Additionally, participants reported their current health status using a visual analog scale (EQ-VAS) that ranged from 0 (indicating the lowest health status) to 100 (indicating the highest health status) points.

Demographic data were also collected, including information on gender, age, BMI, duration of diabetes mellitus (DM), fasting blood sugar value, ethnicity, occupation status, education level, religion, smoking status, type of diabetes, diabetes treatment, presence of DM complications, foot deformities, history of previous amputation, and time elapsed since the last ulcer healed.

2.3. Data Analysis All data were analyzed using SPSS software (version 26.0; IBM Corp., Armonk, NY, USA). The demographic variables were assessed using descriptive statistics (means, standard deviation, frequencies). A mixed model for repeated measures analysis was used to test the differences in quality of life and high-risk level on baseline and the third follow-ups between the two groups. p < 0.05 was chosen as the level of significance

ELIGIBILITY:
Inclusion Criteria:

* Participants have a history of diabetic foot ulcers.
* signed an informed consent

Exclusion Criteria:

* Declined to participate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
The degree of risk of recurrence | up to three months
  The risk level recurrence ulcer tool, INDIFURUTO (Indonesian Diabetic Foot Ulcer Recurrence Assessment Tool), was used to assess the risk level. Subjects were categorized as high risk if they scored less than or equal to 22 points, medium risk if they scored between 23 and 45, and low risk if they scored more than or equal to 46.
Efficacy of prevention strategies | up to three months
  Prevention stratagies is evaluated using INDIFURUTO tool (history of amputation, smoking, serum glucose levels, ankle-brachial index, monofilament test results, and differences in foot skin temperature). Good=INDIFURUTO total score increase than baseline and Poor=INDIFURUTO total score decrease than baseline

SECONDARY OUTCOMES:
Quality of life of DFU's | up to three months
  The European Quality of Life 5 Dimensions 3 Level (EQ-5D-3L) version was used to evaluate participants' quality of life. Level 1 (indicating the best state) to Level 3 (indicating the worst state).
Health status of DFU's | up to three months
  Health status using a visual analog scale (EQ-VAS) that ranged from 0 (indicating the lowest health status) to 100 (indicating the highest health status).

CONTACTS AND LOCATIONS:
Overall Officials: Haryanto Haryanto, Study Chair — ITEKES Muhammadiyah Kalimantan Barat
Locations (1):
- Haryanto Haryanto, Pontianak, West Kalimantan, Indonesia

REFERENCES:
- [Derived] Haryanto H, Sari Y, Panjaitan E, Juminar J, Armstrong D. A Randomized Clinical Trial Study on the Prevention Strategy and Early Detection of Ulcer Recurrence in Patients with Type 2 Diabetes Mellitus Using the Risk of Recurrence Ulcer Tool. Int J Low Extrem Wounds. 2025 Sep;24(3):655-663. doi: 10.1177/15347346241283160. Epub 2024 Oct 21. PMID 39434549